CLINICAL TRIAL: NCT05408559
Title: Prevention of Age-associated Cardiac and Vascular Dysfunction Through Nrf2 Signaling Using the Nutritional Supplement Sulforaphane
Brief Title: Prevention of Age-associated Cardiac and Vascular Dysfunction Using Avmacol ES
Acronym: CardiacAging
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: L22-024
Record Dates: First submitted 2022-03-17; First posted 2022-06-07 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Diastolic Dysfunction; Systolic Dysfunction; Diastolic Heart Failure
Keywords: Sulforaphane; oxidative stress; HFpEF; HFrEF; Arterial function; Muscle function
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — sulforaphane

STUDY DESIGN:
Intervention Model Description: Well trained Nurses of Clinical Research Institute, TTUHSC will receive placebo and test compound from supplier and will dispense them to test subjects.
Who Masked: Participant
Masking Description: These potential subjects will be recruited in a randomized, controlled, double blinded pilot study comparing SFN to placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avmacol ES (Active Comparator): Processed SFN-rich extract will be purchased from Nutramax Laboratories, Inc. 2208 Lakeside Blvd Edgewood, MD 21040. Caplets containing SFN-rich broccoli sprout extracts will be obtained from Nutramax Labs. Study medication will be dispensed in sealed bottles with instructions to keep them in a household freezer. The size of the caplet will be about the size of a 1000 mg Vit C pill (about 2 cm in length). The participants will be dosed, based on weight, in a double-blind fashion with identical appearing placebo or SFN caplets. Participants will be instructed to take a daily dose for 24 weeks based on the participants weight. Two caplets for individuals <100 lb., three caplets for individuals 100-200 lb. and four caplets for individuals >200 lb. SFN (Avmacol Extra Strength) will be prescribed by a study physician, and will be dispensed by the study coordinators at TTUHSC Lubbock. Pill counts will be conducted to demonstrate compliance.
  Interventions: Drug: Sulforaphane
- Placebo (Placebo Comparator): Placebo caplets containing microcrystalline cellulose will be obtained from Nutramax Labs. Study medication will be dispensed in sealed bottles with instructions to keep them in a household freezer. The size of the caplet will be about the size of a 1000 mg Vit C pill (about 2 cm in length). The participants will be dosed, based on weight, in a double-blind fashion with identical appearing placebo or SFN caplets. Participants will be instructed to take a daily dose for 24 weeks based on the participants weight. Two caplets for individuals <100 lb., three caplets for individuals 100-200 lb. and four caplets for individuals >200 lb. Placebo will be prescribed by a study physician, and will be dispensed by the study coordinators at TTUHSC Lubbock. Pill counts will be conducted to demonstrate compliance.
  Interventions: Drug: Sulforaphane

INTERVENTIONS:
Drug: Sulforaphane — Caplets containing SFN-rich broccoli sprout extracts or placebo caplets containing microcrystalline cellulose will be obtained from from Nutramax Labs.
  Other Names: Avmacol Extra Strength

SUMMARY:
Our local IRB approved clinical studies seeking proof of principle for the hypothesis that SFN can be safely administered to humans at doses sufficient to protect age-associated cardiac dysfunctions. Beneficial effects of SFN-therapy will be assessed by Pre- and post-intervention echocardiography, and exercise endurance at 0 and 24 weeks. Peripheral blood cells from treated and control subjects will be compared for mitochondrial respiratory function, oxidative damage, pro-inflammatory cytokines, and expression of antioxidant & anti-electrophile genes.

DETAILED DESCRIPTION:
Study Design: We intend to include 200 individuals (100 men and 100 women, ≥60 years), with a diagnosis of heart failure with preserved ejection fraction (HFpEF) who are able to walk at least 500 feet, to participate in a randomized controlled, double blinded study, with Sulforaphane (SFN) or placebo treatment for 24 weeks. These potential subjects will be recruited in a randomized, controlled, double blinded pilot study comparing SFN to placebo. The study will be conducted at the Texas Tech University Health Sciences Center, and University Medical Center. The trial is approved by our local IRB (IRB NUMBER: L22-024, IRB APPROVAL DATE: 12/14/2021) and will be registered at clinicaltrials.gov. Well trained Nurses of Clinical Research Institute, TTUHSC will receive placebo and test compound from supplier and will dispense them to test subjects.

Sulforaphane and Placebo Information. Processed SFN-rich extract will be purchased from Nutramax Laboratories, Inc. 2208 Lakeside Blvd Edgewood, MD 21040. Caplets containing SFN-rich broccoli sprout extracts or placebo caplets containing microcrystalline cellulose will be obtained from from Nutramax Labs. Study medication will be dispensed in sealed bottles with instructions to keep them in a household freezer. The size of the caplet will be about the size of a 1000 mg Vit C pill (about 2 cm in length). The participants will be dosed, based on weight, in a double-blind fashion with identical appearing placebo or SFN caplets. Participants will be instructed to take a daily dose for 24 weeks based on the participants weight. Two caplets for individuals <100 lb., three caplets for individuals 100-200 lb. and four caplets for individuals >200 lb. SFN (Avmacol Extra Strength) or placebo will be prescribed by a study physician, and will be dispensed by the study coordinators at TTUHSC Lubbock. Pill counts will be conducted to demonstrate compliance.

The study medications will arrive pre-packaged and be stored in a refrigerator freezer in the TTUHSC Clinical Research Institute based on the manufacturer-based guidelines and dispensed to each participant at their baseline visit and at the 12 weeks visit. Patients will be expected to maintain at least an 80% adherence to the medication regimen, in the absence of prohibitive toxicity. Adherence will be monitored through pill counts. Subjects who do not meet 80% compliance when questioned with phone visits and at 12-week pill count, will be instructed on the importance of taking the pills as directed, but if they demonstrate less than 80% compliance on average for more than 2 in person and/or phone study visits, they will be withdrawn from the study, and we will not use their data. If side effects are noted, patient will be asked to notify the study team of the same and will be evaluated within a suitable time frame based on severity of side effects.

SFN is a safe natural isolate. The doses that are used in this study as described above (30mg/caplet) are considered adequate to maintain intended therapeutic drug levels, while maintaining a simple study design without significant concerns for drug toxicity. SFN has been used in several clinical trials from doses ranging from 2-200µmol/day for 2-28 weeks in 25-80 years old subjects without significant side-effect or toxicity (https://clinicaltrials.gov/ct2/results?term=sulforaphane&Search=Search ).

Data Analysis and Statistical Considerations: Data will be analyzed using SPSS 21.0 (for Windows, SPSS Inc., Chicago, IL). Descriptive statistics and correlation analysis will be performed. All results will be expressed as mean±SE. The significance of difference in mean values between groups will be examined using analysis of variance (ANOVA) or, when the ANOVA assumptions are not fulfilled, using the Mann-Whitney (if two groups are to be compared) or Kruskal Wallis (if three or more groups are to be compared) non-parametric test. These tests will be followed by Tukey's HSD test for means or ranks if appropriate (SPSS 21.0). For evaluating changes in cardiac function and LV mass over time, a mixed-design ANOVA, implemented with generalized linear models, will be used. A value of P ≤ 0.05 will be considered statistically significant.

Power analysis: The number of subjects per group is based on previous results from studies using anabolic agents in older adults. The power analysis assuming an equal sample size and variability among the groups, α=0.05, 80% power and 30% expected difference in means, was found to be n=100/group, this allows for an anticipated 10-20% attrition rate.

Study visits/Roles of subjects: Informed consent will be obtained from participants prior to any study procedures. Before and after the intervention, the subjects will be tested at the TTUHSC/UMC Cardiology lab, Lubbock. Subjects will undergo baseline health screening which will include a health status questionnaire (SF-36) which will be repeated at 12 and 24 weeks.

Echocardiography. Echocardiography will be performed at TTUHSC/UMC Cardiology Lab using a commercially available echocardiography unit (Vivid E9, GE, Waukesha, WI, USA) to assess left ventricular (LV) mass, LV systolic and diastolic function as described previously, at Baseline and 24 weeks visits. Speckle tracking echocardiography will be used to assess global longitudinal strain at baseline and its response to treatment. Echocardiography will be performed by registered sonographers and interpreted by a cardiologist with advanced training in echocardiography (level 3 certified). Both the sonographer and the interpreter will be blinded to treatment allocation.

Response to exercise. After resting echocardiogram is performed, all subjects will be subjected to treadmill exercise test using the Bruce protocol (at baseline, 12 and 24 weeks). Tests will be performed in a standard fashion and exercise capacity will be expressed in metabolic equivalents (METS) which are derived from standard published nomograms based on the time on the treadmill. We will also perform the 6 minute walk test on a hard, flat surface at baseline, and 24 weeks to assess functional capacity.

Muscle function. Muscle function will be determined by established strength and endurance tests. These are the treadmill tests above and the hand grip test. Hand grip strength. Hand grip strength will be measured at baseline, 24 weeks using a Jamar hand dynamometer.

Blood samples. Approximately 10 ml of blood will be drawn from the participants before starting SFN (or placebo) at Baseline and 24 weeks using aseptic techniques. Peripheral blood mononuclear cells will be isolated within 4 hours of blood draw from a portion of the blood to analyze the reactive oxygen species formation, markers of oxidative damage, inflammatory signals (CRP, IL-6 and IL-10), mRNA expression levels of Nrf2 target genes and Nrf2/ARE binding. As described:

* Assessment of oxidative damage. Oxidative biomarkers in skeletal muscle, such as 8-oxo-7,8-2'-deoxyguanosine (DNA) and lipid peroxidation (MDA), will be measured by ELISA, spectrophotometry, Western blot analysis and immunohistochemistry, utilizing commercially available kits and appropriate antibodies.
* Determination of antioxidant/anti-electrophile mRNA levels by real-time polymerase chain reaction. Total RNA will be isolated from skeletal muscle and peripheral blood mononuclear cells samples of study participants by the guanidinium thiocyanate method. Complementary DNA will also be prepared using cDNA synthesis kit (Thermo Scientific, Waltham, MA). Real-time polymerase chain reactions (qPCR) will be performed in triplicate on a DNA Engine Opticon 2 Detection System (MJ Research, Waltham, MA) with the SYBR select Master mix from Applied Biosystems (Grand Island, NY).
* The complete blood count (CBC), and CMP tests will be used as a broad screening test. If an adverse event occurs and the study physician thinks it is necessary for the patient's safety, these tests will be performed to determine an individual's general health status.

Arterial function. Pulse wave velocity is a marker of endothelial function and predicts cardiovascular events. Subjects will undergo noninvasive arterial function testing at Baseline and 24 weeks using an FDA-approved device (Sphygmocor XCEL) at TTUHSC/UMC cardiology lab.

Study Population We will recruit up to 200 volunteers (100 men and 100 women), ≥65 years, with diagnosis of HFpEF (HF symptoms with a normal EF). Participants will be recruited from the Cardiology Clinic and by the use of the Clinical Research Institute's volunteer database, advertisements, notices, and/or media. Examples include IRB approved flyers posted in public settings at TTUHSC, the TTUHSC Cardiology Clinic, and newspaper advertisement. All advertisements and recruitment materials will be IRB approved. Anyone contacting the research team in response to an advertisement/flyer will be pre-screened for study eligibility. We will consent volunteers to participate in a randomized controlled, double blinded study, with SFN or placebo treatment for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Diagnosis of HFpEF (HF symptoms with a normal EF (>/=50 %)
* Ability to walk more than 500 feet (by self-report)
* Willing to avoid taking all over the counter antioxidant phytochemical supplements (vegetable or fruit-containing supplement pills) during the study

Exclusion Criteria:

* Inability to provide informed consent
* Diagnosis of active cancer
* Inability to read and understand the SF-36 in English
* Participants using over the counter antioxidant supplements
* Participants with pulmonary or other issues which restrict walking capacity
* On oxygen therapy

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
cardiac function | 0 week
  1. LV ejection fraction at baseline and 24 weeks
  2. Left ventricular global longitudinal strain at baseline and 24 weeks
  3. Left ventricular diastolic function at baseline and 24 weeks
cardiac function | 24 week
  1. LV ejection fraction at baseline and 24 weeks
  2. Left ventricular global longitudinal strain at baseline and 24 weeks
  3. Left ventricular diastolic function at baseline and 24 weeks
Functional Capacity | 0 week
  Exercise capacity in METS at baseline and 24 weeks
Functional Capacity | 24 week
  Exercise capacity in METS at baseline and 24 weeks

SECONDARY OUTCOMES:
Muscle Function | 0 week
  Muscle function will be determined by established strength and endurance tests
Muscle Function | 24 week
  Muscle function will be determined by established strength and endurance tests
Hand grip test | 0 week
  Determined using a Jamar hand dynamometer
Hand grip test | 24 week
  Determined using a Jamar hand dynamometer

OTHER OUTCOMES:
DNA damage, CBC, Oxidative stress | 0 week
  Measured in Peripheral Blood cells
DNA damage, CBC, Oxidative stress | 24 weeks
  Measured in Peripheral Blood cells

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University Health Sciences Center (TTUHSC), Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Results of this study may be used for presentations, posters, or publications. The publications will not contain any identifiable information that could be linked to a participant.